CLINICAL TRIAL: NCT05469555
Title: Exploring the Effect of Azithromycin on Oesophageal Motility and Respiratory Symptoms in Patients With Chronic Respiratory Disease: a Prospective Observational Study
Brief Title: Azithromycin and Oesophageal Function in Respiratory Disease
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 315000
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cough; Asthma; Copd; ILD
MeSH Terms: conditions — Cough; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: High Resolution Oesophageal Manometry — High Resolution Oesophageal manometry assesses how well the muscles of the oesophagus are working when you swallow. It also checks the relaxation of the valves at the top and bottom of the oesophagus.

SUMMARY:
Symptoms such as cough, wheeze, and breathlessness are among the most common reasons for general practitioner or emergency department visits in the UK. Such symptoms have a profound impact on patients' ability to live a fulfilled life, often rendering people unable to work and socialise.

Azithromycin (a type of antibiotic) improves symptoms and reduces flare-ups of diseases such as asthma and chronic obstructive pulmonary disease (COPD). The reason why it works is unclear. Many people believe that it either decreases the number of bacteria in the lungs or reduces inflammation in the lungs and the upper airways. Neither theory is proven. Another possible mechanism that has been much less studied is that Azithromycin encourages the body to move food and fluid through the gut more quickly, thus preventing reflux and aspiration of small food particles and stomach acid. It has been shown that lung damage can occur when gut contents enter the airways, which may contribute chronic lung disease patients' symptoms

In this study the investigators will test the effect of azithromycin on the gut in patients with chronic lung diseases. The investigators will measure the strength of a patients swallow by measuring the pressures in their gullet, using high-resolution oesophageal manometry (HROM), before and after treatment, in people being started on azithromycin as part of their routine care. The investigators will also measure the effect that azithromycin has on their symptoms and observe whether there is a relationship between the strength of their swallow and their symptoms.

At the end of this study, the investigators hope to better understand the way in which azithromycin helps to improve the symptoms of patients with chronic lung diseases. The investigators also hope to open the door to investigate the effect of other drugs that improve gut function in patients with chronic lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥18 years.
* Have a diagnosis of chronic respiratory disease (COPD, asthma, interstitial lung disease, chronic cough, cystic fibrosis, and/or bronchiectasis) confirmed by a respiratory consultant.
* Exhibit symptoms consistent with airway reflux, demonstrated by a score ≥14 on the Hull Airways Reflux Questionnaire
* Are being initiated on azithromycin as part of routine clinical care, as judged by their usual respiratory clinician. This will include all common treatment regimes, 250mg once daily, 250mg three times per week, and 500mg three time per week.
* Are willing and able to consent to all study procedures.

Exclusion Criteria:

* Previous treatment with long-term macrolides in the past 3 months.
* Unable to be investigated with HROM due to contraindications such as anatomical abnormalities or diseases of the oesophagus or unwilling/ unable to be investigated with HROM based on the clinical judgement of the investigators due to severity of lung disease.
* Have another cardiorespiratory cause for their symptoms (such as heart failure or lung cancer).
* Women of child bearing potential not using effective means of contraception.
* Are unable or unwilling to consent to or complete the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic respiratory disease whose normal respiratory physician is considering initiating azithromycin therapy for.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Eligibility to consent ratio | 1 year
  The ratio of participants deemed eligible to participate in the study to the number of those who provide consent to take part
Recruitment rate | 1 year
  The number of participants successfully recruited per month
Participant retention to follow-up | 1 year
  The proportion of those participants who consent to take part that compete all study measures to follow-up
Acceptability of assessment | 1 year
  Quantify the proportion of participants who judge the study investigations, principally HROM, to be acceptable.

SECONDARY OUTCOMES:
Distal Contractile Integrity | 1 month
  To evaluate the effect of azithromycin on the contraction vigour and swallow coordination. This will be evaluated by investigating patients with HROM before and 1 month after initiation of azithromycin as part of routine clinical care. Measured in mmHg/sec/cm.
Lower Oesophageal Sphincter Pressure | 1 month
  To evaluate the effect of azithromycin on the pressure of the lower oesophageal sphincter as measured by HROM. This will be evaluated by investigating patients with HROM before and 1 month after initiation of azithromycin as part of routine clinical care. Measured in mmHg.
Distal Latency | 1 month
  To evaluate the effect of azithromycin on the timeframe of the wave from the beginning of the swallow to an inflection of the peristaltic axis, as measured by HROM. This will be evaluated by investigating patients with HROM before and 1 month after initiation of azithromycin as part of routine clinical care. Measured in seconds.
Integrated Relaxation Pressure. | 1 month
  To evaluate the effect of azithromycin on the oeosphageal pressure topography metric that is used for assessing the adequacy of oesophageogastric junction relaxation, as measured by HROM. This will be evaluated by investigating patients with HROM before and 1 month after initiation of azithromycin as part of routine clinical care. Measured in seconds.
Chicago Classification | 1 month
  A composite classification based on all HROM measurements. We will be using the current version 4.0.
Hull Airway Reflux questionnaire | 1 month
  A validated tool for assessing symptoms of reflux. A likert scale questionnaire. Scored out of 70 with higher score representing worse symptoms.
Breathlessness, cough, and sputum scale | 1 month
  A validated tool for assessing symptom burden. A 5-point likert scale that is scored out of 12. A higher score representing worse symptoms.
MRC dyspnoea scale | 1 month
  A validated tool for measuring breathlessness. It is scored out out of 5 with a higher score representing worse symptoms.
Visual analogue scale - cough severity | 1 month
  A visual scale of 100mm in length. Participants will mark on the scale from 0-100 how bad their cough is currently with 100mm representing worst cough imaginable.
COPD Assessment test (COPD patients only) | 1 month
  An 8 item questionnaire which quantifies the symptom burden participants with COPD and how it impacts their life. Scored out of 40, with a higher score signifying worse control.
Asthma control questionnaire (asthma patients only) | 1 month
  An 7 item questionnaire which quantifies the symptom burden participants with asthma and how it impacts their life. Scored 5-25 - a score of 5 is very poorly controlled asthma and a score of 25 is very well controlled asthma.
Numerical rating scale - breathlessness severity | 1 month
  A horizontally arranged scale numbered 0-10 with 0 representing no breathlessness and 10 representing the worst breathlessness imaginable
Leicester Cough Questionnaire | 1 month
  A 19-item questionnaire with a 7-point Likert scale used to assess the impact of cough on physical, social, and psychological welfare of the patient. It is scored out of 133 with a higher score representing better health.
St. George's Respiratory Questionnaire | 1 month
  A 50-item questionnaire which assess impact of overall health, daily life, and well-being in patients with obstructive airways disease. Scores range from 0-100, with higher scores indicating more limitations.
King's Brief Interstitial Lung Disease Questionnaire (ILD Patients only) | 1 month
  A 15-item 7-point Likert scale questionnaire aimed to measure the impact of ILD on quality of life and health status. It is scored out of 100, with 100 representing the best health status.
Relationship between oesophageal motility and symptoms | 1 month
  The change in oesophageal functioning and presence of respiratory symptoms will be examined in each participant. The relationship between these two parameters will then be examined using statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, Yorkshrie, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sykes DL, Brindle K, Menon R, Hart SP, Nielsen J, Jackson W, Gallagher J, Kirton E, Zhang M, Morice AH, Crooks MG. Azithromycin and oesophageal motility in chronic respiratory disease: a feasibility study. Ther Adv Respir Dis. 2025 Jan-Dec;19:17534666251360065. doi: 10.1177/17534666251360065. Epub 2025 Jul 29. PMID 40734318